CLINICAL TRIAL: NCT03223909
Title: Efficacy and Safety of the Ophthalmic Solution PRO-087 Versus Systane ® Ultra and Systane ® Ultra Preservative Free on Tear Film Dysfunction Syndrome From Mild to Moderate
Brief Title: Efficacy and Safety of the Ophthalmic Solution PRO-087 Versus Systane ® Ultra and Ultra Preservative Free (087LATAMFIV)
Acronym: 087LATAMFIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH087-0415/IV
Record Dates: First submitted 2017-06-22; First posted 2017-07-21 (Actual); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Syndrome
Keywords: dry eye; Chondroitin sulfate; Ocular lubricants
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Chondroitin Sulfates; Hyaluronic Acid; polyethylene glycol 400; Propylene Glycol

STUDY DESIGN:
Intervention Model Description: Controlled, double-blind, randomized, clinical trial comparing the safety and efficacy parameters between a group of subjects with a diagnose of mild to moderate tear film dysfunction syndrome under a regimen of ophthalmic solution lubricant drops PRO-087 versus subject under Systane® Ultra or Systane® Ultra preservative free, with the same diagnosis, with a follow-up of 90 days.
Who Masked: Participant, Investigator
Masking Description: The double-blind study is a procedure in which the patient and the treating doctor ignore to which intervention group the study patient was assigned. To achieve the blinding of both the drug in research and both comparator drugs, these will be labeled in the same way (masking). Besides the figure of an unblinded pharmacist, who is responsible for the delivery of the medication to the patient, will be added. Blinding codes are protected by an outsider appointed by the study sponsor. The codes are also available in the research center (fully sealed), so that they can be consulted by the investigator in case a subject presents a serious adverse event, prior authorization from the study sponsor; the blinding also continues rigorous during the data analysis and interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRO-087 PF (Experimental): Preservative free (PF) PRO-087 ophthalmic solution. Dropper bottle. Multidose 1 drop every 4 hours for 90 days.
  Interventions: Drug: PRO-087
- Systane Ultra (Active Comparator): Systane Ultra ophthalmic solution, Dropper bottle, Multidose.
  1 drop every 4 hours for 90 days.
  Interventions: Drug: Systane Ultra
- Systane Ultra PF (Active Comparator): Systane Ultra, preservative free ophthalmic solution, single-use vials.
  1 drop every 4 hours for 90 days.
  Interventions: Drug: Systane Ultra Preservative Free

INTERVENTIONS:
Drug: PRO-087 — 0.1% sodium hyaluronate, free-preservative 0.18% chondroitin sulphate
  Other Names: Chondroitin sulfate; sodium hyaluronate
  Arms: PRO-087 PF
Drug: Systane Ultra — Is a sterile solution containing polyethylene glycol 400, propylene glycol, hydroxypropyl-guar, sorbitol, aminomethylpropanol, boric acid, potassium chloride, sodium chloride and POLYQUAD® (poly-hydronium chloride) 0.001% as preservative.
  Other Names: polyethylene glycol 400, propylene glycol
  Arms: Systane Ultra
Drug: Systane Ultra Preservative Free — Polyethylene Glycol 400 0.4%Lubricant, Propylene Glycol 0.3% Lubricant,
  Other Names: Polyethylene Glycol 400 0.4%, Propylene Glycol 0.3%
  Arms: Systane Ultra PF

SUMMARY:
Efficacy and Safety of the Ophthalmic Solution PRO-087 versus Systane ® Ultra and Systane ® Ultra Preservative Free on the Tear Film Dysfunction Syndrome from Mild to Moderate Clinical trial To evaluate the effectiveness of preservative-free ophthalmic formulation PRO-087 (by Laboratorios Sophia, S.A. de C.V.) to restore the anatomical and physiological characteristics of the ocular surface, as well as its distribution and the characteristics of the mild to moderate tear film dysfunction syndrome compared to Systane ® Ultra and Ultra Systane ® preservative free (by Laboratorios Alcon, S.A. de C.V.).

Controlled, randomized, double-blind, masked clinical study, comparing the safety and efficacy of preservative-free PR0-087 vs Systane Ultra with preservative and Systane Ultra preservative free, in subjects with mild to moderate tear film dysfunction syndrome, for a period of 90 days plus 15 days of remote surveillance, in which one of the three agents will be administered (PR0-087, Systane® Ultra or Systane® Ultra preservative free) with a q.i.d. dosage. in both eyes, with regular follow-up visits (5 overall).

Best-corrected visual acuity Intraocular pressure Ocular surface Anterior segment examination Posterior segment examination Tear film break-up time Schirmer test Corneal epithelization Goblet cells count Adverse events Subjects with a clinical diagnosis of mild to moderate tear film dysfunction syndrome between 18 and 90 years old, without concomitant eye diseases nor requiring different treatments of any of the three interventions in this study They will be randomized in 3 groups where PRO-087, Systane® Ultra o Systane® Ultra preservative free will be administered.

DETAILED DESCRIPTION:
Design Controlled, double-blind, randomized, clinical trial comparing the safety and efficacy parameters between a group of subjects with a diagnose of mild to moderate tear film dysfunction syndrome under a regimen of ophthalmic solution lubricant drops PRO-087 versus subject under Systane® Ultra or Systane® Ultra preservative free, with the same diagnosis, with a follow-up of 90 days

MAIN OBJECTIVE:

To evaluate the effectiveness of preservative-free ophthalmic formulation PRO-087 (by Laboratorios Sophia, S.A. de C.V.) to restore the anatomical and physiological characteristics of the ocular surface, as well as its distribution and the characteristics of the mild to moderate tear film dysfunction syndrome compared to Systane ® Ultra and Ultra Systane ® preservative free (by Laboratorios Alcon, S.A. de C.V.).

SPECIFIC OBJECTIVES:

To evaluate the safety of the preservative-free ophthalmic formulation PRO-087 (by Laboratorios Sophia, S.A. de C.V.) on the corneal and conjunctival epithelium, intraocular pressure, and structures of anterior and posterior segment in patients with tear film dysfunction syndrome from mild to moderate.

To determine the correlation between improvement of clinical status and perceived improvement of symptoms of each participant in each study group.

To compare the qualitative and quantitative histological status of the ocular surface before and after the pharmacological intervention in each study group to determine the evolution under the intervention of PRO-087.

To evaluate the quantitative rating of tear film production by the Schirmer Test throughout the study.

To qualitatively assess the tear film production by measuring the tear film break-up time stained with fluorescein and cobalt filter.

Blinding:

The double-blind study is a procedure in which the patient and the treating doctor ignore to which intervention group the study patient was assigned. To achieve the blinding of both the drug in research and both comparator drugs, these will be labeled in the same way (masking). Besides the figure of an unblinded pharmacist, who is responsible for the delivery of the medication to the patient, will be added. Blinding codes are protected by an outsider appointed by the study sponsor. The codes are also available in the research center (fully sealed), so that they can be consulted by the investigator in case a subject presents a serious adverse event, prior authorization from the study sponsor; the blinding also continues rigorous during the data analysis and interpretation.

patients with tear film dysfunction, classified as mild to moderate, will be included and randomized into 3 groups; the first being treated with PRO-087 ophthalmic solution, the second with Systane® Ultra ophthalmic solution, and the third with ophthalmic solution Systane® Ultra preservative free.

Pharmacological Intervention

The pharmacological intervention will be the instillation of the ophthalmic solution in the bottom of the conjunctival sac during the waking period, in any of the following study groups:

1. Preservative free PRO-087 ophthalmic solution. Dropper bottle. Multidose 1 drop every 4 hours for 90 days.
2. Systane® Ultra ophthalmic solution. Dropper bottle. Multidose. 1 drop every 4 hours for 90 days.
3. Systane ® Ultra preservative free ophthalmic solution. Single-use vials. 1 drop every 4 hours for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* >18 to < 90 years old
* Both sexes
* Mild to moderate tear film dysfunction clinical diagnose
* Mild to moderate clinical stage of the disease

  * TBUT > 5 sec. and < 10 sec.
  * Schirmer: > 4 mm and < 14 mm
  * OSDI < 30 points
  * Corneal staining < grade III on the Oxford scale
* Availability to go to each revision when indicated.

Exclusion Criteria:

General Criteria

1. Subjects with topical and/or systemic medication or mechanical devices that interfere determinedly on the results of the study (such as topical immunomodulators, punctal plugs, corticosteroids, preservative artificial tears, contact lenses).
2. Subjects (females) with active sexual life that do not use a contraceptive method.
3. Female subjects who are pregnant or lactating
4. Female subjects with a positive urine pregnancy test
5. Positive drug addictions* (verbal interrogatory)
6. Subjects who have participated on any other research clinical trials on the last 40 days
7. Subjects legal or mentally disabled to give an informed consent for participating on this study
8. Subjects who can't comply with the appointments or with every protocol requirement.

Criteria related with ophthalmic ailments

1. Serious tear film dysfunction syndrome TBUT < 5 s Schirmer: < 4 mm OSDI > 30 pints Corneal staining > grade III on the Oxford scale
2. Non perforated corneal ulcer
3. Perforated corneal ulcer
4. Autoimmune corneal ulcer
5. Ocular surface scarring diseases
6. Ocular surface or annexes metaplastic lesions
7. Fibro vascular proliferation lesions on the conjunctival and/or corneal surface (i.e.: pterygium)
8. Concomitant chronic inflammatory diseases on any ocular structure
9. Acute or infectious inflammatory disease
10. Corneal disease potentially requiring a treatment during the following 3 months
11. Use of topical or systemic drug products classified as forbidden
12. Ocular surgical procedures 3 months before the protocol inclusion
13. Treatments or procedures indicated on the tear film dysfunction treatment, as punctal silicone plugs.
14. Posterior segment diseases requiring a treatment or threatening the visual prognosis
15. Retinal diseases potentially requiring treatment during the following 3 months
16. History of penetrating keratoplasty.
17. Soft or hard contact lenses use during the last month from inclusion day

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2016-10-13 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Fernando Rodriguez Sixtos Higuera, Irapuato, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No
For security and laws implemented by the regulatory entity can not share personal data of research subjects.

RESULTS

PARTICIPANT FLOW:
Groups:
- Systane Ultra: Systane Ultra ophthalmic solution, Dropper bottle, Multidose.
  1 drop every 4 hours for 90 days.
  Systane Ultra: Is a sterile solution containing polyethylene glycol 400, propylene glycol, hydroxypropyl-guar, sorbitol, aminomethylpropanol, boric acid, potassium chloride, sodium chloride and POLYQUAD® (poly-hydronium chloride) 0.001% as preservative.
- Systane Ultra PF: Systane Ultra, preservative free ophthalmic solution, single-use vials.
  1 drop every 4 hours for 90 days.
  Systane Ultra Preservative Free: Polyethylene Glycol 400 0.4%Lubricant, Propylene Glycol 0.3% Lubricant,
Period: Overall Study
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Started | 120 | 109 | 97
Completed | 72 | 64 | 81
Not Completed | 48 | 45 | 16
Not completed — Protocol Violation | 48 | 45 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF | Total
Number analyzed (Participants) | 72 | 64 | 81 | 217
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (15.3) | 55.0 (17.6) | 51.9 (16.2) | 54.2 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 46 | 63 | 161
  Male | 20 | 18 | 18 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 72 | 64 | 81 | 217
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity
Description: Best-corrected visual acuity
Time Frame: Change from Baseline visual acuity at 90 days
Population: the statistical analysis was carried out by intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
LogMAR
  Base Line | 0.187 (0.25) | 0.215 (0.26) | 0.219 (0.23)
  Final Visit | 0.172 (0.24) | 0.187 (0.24) | 0.176 (0.21)
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20% Statistical analysis of groups in the baseline visit versus final visit; p = 0.080, ANOVA
Statistical Analysis 2: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20% Statistical analysis between groups in the final visit; p = 0.848, ANOVA

2. Secondary Outcome: Corneal Epithelization Defects With Rose of Bengal
Description: Percentage of the damaged epithelium of the ocular surface, reduction of staining according to the oxford scale.
Time Frame: Final Visit (day 90)
Population: the statistical analysis was carried out by intention to treat
Measure: Number; unit: percentage of defects
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
percentage of defects
  Normal (0) | 80.6 | 73.4 | 77.8
  Very mild (1) | 18.1 | 25 | 19.1
  Mild (2) | 1.4 | 1.6 | 3.1
  Moderate (3) | 0 | 0 | 0
  Severe (4) | 0 | 0 | 0
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20%; p = 0.468, Chi-squared, Corrected

3. Secondary Outcome: Tear Film Break-up Time (TBUT)
Description: Tear breakup time (TBUT) is a clinical test used to assess for evaporative dry eye disease. To measure TBUT, fluorescein is instilled into the patient's tear film and the patient is asked not to blink while the tear film is observed under a broad beam of cobalt blue illumination. The TBUT is recorded as the number of seconds that elapse between the last blink and the appearance of the first dry spot in the tear film, as seen in this progression of these slit lamps photos over time. A TBUT under 10 seconds is considered abnormal
Time Frame: Base line and Final Visit (day 90)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
seconds
  Base Line | 7.08 (1.01) | 7.10 (1.01) | 7.10 (1.01)
  Final visit | 8.28 (2.3) | 8.46 (2.6) | 8.52 (2.2)
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — population analysis was per protocol; p = 0.0001, ANOVA
Statistical Analysis 2: Comparison: PRO-087 PF vs Systane Ultra; Test type: Non-Inferiority — population analysis was per protocol; p = 0.650, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Schirmer Test
Description: Schirmer's test determines whether the eye produces enough tears to keep it moist. This test is used when a person experiences very dry eyes or excessive watering of the eyes. It poses no risk to the subject. A negative (more than 10 mm of moisture on the filter paper in 5 minutes) test result is normal. Both eyes normally secrete the same amount of tears.
Time Frame: Base line and Final Visit (day 90)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
mm
  basal visit (day 1) | 9.48 (2.5) | 9.05 (2.7) | 9.25 (2.7)
  Final Visit | 10.19 (4.2) | 12.21 (4.5) | 12.16 (5.6)
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra; Test type: Non-Inferiority — It was considered as not inferior when the treatments did not present differences greater than 20% Statistical analysis of Humylub® Ofteno (PRO-087) versus Systane® Ultra PF at the final visit; p = 0.003, ANOVA
Statistical Analysis 2: Comparison: PRO-087 PF vs Systane Ultra PF; Test type: Non-Inferiority — [test comment as in outcome 4, analysis 1]; p = 0.003, ANOVA

5. Secondary Outcome: Adverse Events
Description: Presence of adverse events modifying some of the abovementioned criteria or others, evaluated as serious.
Time Frame: 90 days
Population: Statistical analysis was performed by protocol (PP)
Measure: Number; unit: percentage of adverse events
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 120 | 109 | 97
percentage of adverse events | 19.2 | 21.1 | 20.6
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — the statistical analysis was carried out by intention to treat It was considered as not inferior when the treatments did not present differences greater than 20%; p = 0.930, Chi-squared

6. Secondary Outcome: Ocular Surface Disease Index (OSDI)
Description: The OSDI, which was created to order to quickly assess the symptoms of ocular irritation in dry eye disease and how they affect functioning related to vision. This 12-item questionnaire assesses dry eye symptoms and the effects it has on vision-related function in the past of the patient's life. The questionnaire has 3 subscales: ocular symptoms, vision-related function, and environmental triggers. Patients rate their responses on a 0 to 4 scale with 0 corresponding to "none of the time" and 4 corresponding to "all of the time." A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Time Frame: Change from Baseline OSDI at 90 days
Population: The statistical analysis was carried out by intention to treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
score on a scale
  Base Line | 16.59 (7.3) | 15.74 (7.0) | 16.31 (7.7)
  Final Visit | 5.99 (8.2) | 7.47 (8.8) | 6.32 (7.7)
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20%; p = 0.548, ANOVA

7. Secondary Outcome: Goblet Cells Population
Description: Increase of 20% from baseline
Time Frame: Change from Baseline Goblet cells population at 90 days
Population: the statistical analysis was carried out by intention to treat
Measure: Mean (Standard Deviation); unit: cells/mm^2
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
cells/mm^2
  Base Line | 341.2 (136.9) | 338.5 (150.6) | 327.4 (146.8)
  Final Visit | 447.3 (173.4) | 413.5 (157.7) | 442.6 (147.2)
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20%; p = 0.170, ANOVA

8. Secondary Outcome: Corneal Epithelization Defects With Fluorescein
Description: Percentage of the damaged epithelium of the ocular surface, reduction of staining according to the oxford scale.
Time Frame: Final Visit (day 90)
Population: the statistical analysis was carried out by intention to treat
Measure: Number; unit: percentage of defects
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
Number analyzed (Participants) | 72 | 64 | 81
percentage of defects
  Normal (0) | 52.8 | 53.1 | 53.7
  Very mild (1) | 36.8 | 36.7 | 10.4
  Mild (2) | 10.4 | 9.4 | 15.4
  Moderate (3) | 0 | 0 | 2.5
  Severe (4) | 0 | 0.8 | 0
Statistical Analysis 1: Comparison: PRO-087 PF vs Systane Ultra vs Systane Ultra PF; Test type: Non-Inferiority — it was considered as not inferior when the treatments did not present differences greater than 20%; p = 0.085, Chi-squared, Corrected

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and recorded throughout the study, an average of 2 years, since october 2016 to october 2018.
Arm/Group | PRO-087 PF | Systane Ultra | Systane Ultra PF
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/109 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/109 | 0/97
Other Adverse Events (participants affected / at risk) | 24/120 | 29/109 | 19/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-087 PF (N=120) | Systane Ultra (N=109) | Systane Ultra PF (N=97)
bacterial conjunctivitis (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
enteroviric gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Defect of the corneal epithelium (Eye disorders) | 6 (6) | 6 (6) | 4 (4)
Bacterial urinary infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Episodes of aggravated nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faringoamigdalitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Urethritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Bacterial gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (General disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic conjunctivitis (Eye disorders) | 1 (1) | 4 (4) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid spasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Nuisance in the area of application (General disorders) | 1 (1) | 0 (0) | 0 (0)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Flexo-extension injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
flu (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Feeling of burning (Eye disorders) | 2 (2) | 1 (1) | 2 (2)
Blurry vision (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Red eye (Eye disorders) | 1 (1) | 1 (1) | 3 (3)
Prurito en el ojo (Eye disorders) | 3 (3) | 3 (3) | 2 (2)
Light fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tearing (Eye disorders) | 4 (4) | 0 (0) | 2 (2)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis of the finger (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Foreign body sensation in the eyes (Eye disorders) | 1 (1) | 2 (2) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Allergy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
IPs may not share, disclose or partially or completely publish the information of this research in order to request and receive written approval from the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT03223909/Prot_SAP_000.pdf